CLINICAL TRIAL: NCT03348787
Title: Behavioral and Cognitive Therapies for Auditory Hallucination Management: Effectiveness and Analysis of Change Processes Involved With Hallucinations in a Population Suffering From Chronic Psychosis
Brief Title: Behavioral and Cognitive Therapies for Auditory Hallucination Management
Acronym: AcceptVoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0159; 2017-A01929-44 (Registry Identifier: French ANSM register)
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Chronic Psychosis
Keywords: Behavioral and Cognitive Therapies
MeSH Terms: conditions — Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral and Cognitive Therapies (Experimental): Chronic psychotic patients will have Behavioral and Cognitive Therapies
  Interventions: Behavioral: Behavioral and Cognitive Therapies

INTERVENTIONS:
Behavioral: Behavioral and Cognitive Therapies — Group intervention of 6 weekly sessions of one hour and 30 minutes based on the psychoeducational therapeutic principles and CBT type 3 wave "Accept Voices" applied to HAV

SUMMARY:
The present study wants to evaluate the efficacy of a short psychoeducational type group intervention and Cognitive behavioral therapy (CBT) 3rd wave on the severity of hallucinatory Acoustico-Verbal (HAV) symptomatology in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic disorders, schizo-affective disorders
* Suffering from persistent HAV
* No change in symptomatology for 3 months.
* No anticipated change in antipsychotic treatment (anti-hallucinatory): olanzapine, risperidone, amisulpride, quetiapine, aripiprazole, loxapine, haloperidol, clopixol, modecate, nozinan, cyamemazine, piportil, clozapine
* Major patient, or major incompetent.

Exclusion Criteria:

* Mental retardation
* Subject participating in another search including an exclusion period still in progress at pre-inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
intensity HAV symptoms | Baseline and one week after the last session
  Difference between the Psychotic Symptom Rating Scales (PSYRATS) on HAV symptom score administered before the first therapeutic group session and the PSYRATS symptom score administered 1 week after the last group session. The PSYRATS Scales measure dimensions of hallucinations and delusions.

SECONDARY OUTCOMES:
Effect over time | Until 12 months after the last session
  Difference between the PSYRATS score given 1 week before the first session, and the PSYRATS score administered one week after the last session and then at 6 weeks, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Bourcier, PhD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - Lannemezan Hospital, Lannemezan
  - Lavaur Hospital, Lavaur
  - Sainte-Marie de Rodez Hospital, Rodez
  - Ariège-Couserans Hospital, Saint-Lizier
  - Gérard Marchand Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No